CLINICAL TRIAL: NCT03863444
Title: I-Yuan Yen, Registered Nurse Department of Nursing, National Taiwan University Hospital
Brief Title: Effects of Prenatal Preparation Education on First-time Parents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201810089RINA
Record Dates: First submitted 2019-02-24; First posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Parenting; Partner, Domestic
Keywords: First-time Parents; Prenatal Preparation Education; Partner Support

STUDY DESIGN:
Intervention Model Description: The study subjects will be divided into the experimental group and control group. In order to avoid the contamination between the control group and the experimental group due to the simultaneous empty space and information sharing, the control group will be recruited in the study in the first two months. After control group recruitment, we will recruit the intervention group and provide prenatal education.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Routine Care
  Interventions: Other: Routine care
- Intervention Group (Experimental): Routine Care + Prenatal Preparation Education
  Interventions: Other: Prenatal Preparation Education; Other: Routine care

INTERVENTIONS:
Other: Prenatal Preparation Education — Intervention, provided by researchers, includes video, counseling, and skill practices. Video contains (1) Newborn Reaction, including rooting reflex, correct latch-on posture, assuring newborn having enough milk intakes; (2) Newborn Care, including holding, dipper-changing, clothes-changing, and swaddle the newborn; and (3) Partner Support, including the importance of partner support and the content how partner provide support to the postpartum women. After watching the video, the researcher will provide participants counseling, and then each pair of participants will have skill practice.
  Arms: Intervention Group
Other: Routine care — Routine care, provided by clinic nurses, includes antenatal breastfeeding education (i.e., providing education sheet, explaining the benefits and importance of breastfeeding, exclusive breastfeeding for six months, responsive breastfeeding, maintaining milk production, immediately skin-to-skin touch after delivery, and room-in) and demonstration of newborn care (i.e., newborns holding posture, breastfeeding holding posture, and newborn latch-on posture) by pictures and baby models.

SUMMARY:
Background: In 2001, the National Health Service of the Ministry of Health and Welfare promoted breastfeeding by adopting the ten measures of successful breastfeeding. However, there is still much room for improvement in Taiwan's continued breastfeeding rate. Currently, although the breastfeeding education is given since pregnancy, the postpartum women were still suffering from baby's and themselves demands, such as unfamiliar with breastfeeding skills, fatigue, discomfort. When the baby is crying, I don't know how to comfort, and I need help from others. The nursing staff cannot provide immediate assistance due to busy clinical work. It showed that it is very important to include the partners to provide assistance and support to postpartum women. The prenatal education for partners is the opportunity to elevate the partners' ability of baby care and support to mothers.

Purpose: The purpose of this study is to explore whether different prenatal education courses increase the ability of prospective parents to breastfeed, infant care, and support, thereby improving the preparation and quality of life in the early postpartum period, reducing the incidence of postpartum depression, promoting the parenting of newborns, and Attachment Study design: This study adopts a class of experimental design, the study recruited pregnant women 35 to 39 weeks of primipara and their spouses, the study subjects were divided into experimental group and control group, calculated by G*Power software, alpha is set as 0.05 while power as 0.8. It should be 51 pair of parents in two groups in the third time point. Considering the possible attrition, the investigators will recruit 80 pairs of the experimental group and the control group, respectively. Data collection was conducted on the structured questionnaire on the prenatal, early postpartum, and one month postpartum to explore the effectiveness of different prenatal education courses for primiparas and their partners.

Expected outcome: The prenatal education is expected to elevate the partners' ability of baby care and support to mothers in early postpartum, to decrease postpartum blue, and to promote the attachment between parents and newborns. The results of the questionnaire will be analyzed using descriptive statistics and inferential statistical analysis using the suite software SPSS 15.0 for Windows.

DETAILED DESCRIPTION:
This study adopts a quasi-experimental design. Eligible subjects are pregnant women 35 to 39 weeks of primipara and their spouses. Specifically, inclusion criteria are (1) gestational age 35 to 39 weeks, (2) adults, (3) primipara and their spouses, (4) having routine prenatal visits and plan to have birth in the medical center, (5) able to communicate with Mandarin or Taiwanese, and (6) willing to participate in this study and give written inform-consent forms. Exclusion criteria are (1) having fetus with abnormality, (2) high-risk pregnancy, and (3) cannot room-in due to newborn's medical conditions. Participants would be assessed on the time points of recruitment (T1), early postpartum during hospitalization (T2), and one-month postpartum (T3).

Before conducting this study, the institutional review board (IRB) has approved this study. The research staffs will approach potential participants during their prenatal visits and invite them to participate in the study. Potential participants would be informed of the study purposes, interventions (routine care for control group, routine care plus intervention for intervention group), and interview contents. After written consent is obtained, the interventions will be arranged. In order to control the quality of data collection, the investigators will train the research assistants. Research training will include ethical concerns about collection of research data, methods of approaching eligible subjects, interviewing techniques, and pilot testing of data collection. The training will provide research assistants by the PI and Co-PI of this study.

ELIGIBILITY:
Inclusion Criteria:

* (1) gestational age 35 to 39 weeks
* (2) adults
* (3) primipara and their spouses
* (4) having routine prenatal visits and plan to have the birth in the medical center
* (5) able to communicate with Mandarin or Taiwanese
* (6) willing to participate in this study and give written inform-consent forms

Exclusion Criteria:

* (1) having fetus with abnormality
* (2) high-risk pregnancy
* (3) cannot room-in due to newborn's medical conditions

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2019-02-25 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Iowa Infant Feeding Attitude Scale (IIFAS) | Parents will be assessed the change among Gestational Week 35~39 (T1), postpartum 3~5 days (T2), and postpartum 1 month (T3).
  The Iowa Infant Feeding Attitude Scale (IIFAS) measured the parents' attitude toward infant feeding with 17 Likert's scale items (Ho & McGrath, 2011). Each item scored from 1 to 5 (1 = strongly disagree, 5 = strongly agree). Items 1, 2, 4, 6, 8, 10, 11, 14, and 17 will be reversed code. The higher score indicated the higher intention to choose breastfeeding; lower scores indicated the intention to choose formula feeding. Cronbach's alpha is 0.75.
Changes of Breastfeeding Self-Efficacy Scale-Short Form (BSES-SF) | Parents will be assessed the change among Gestational Week 35~39 (T1), postpartum 3~5 days (T2), and postpartum 1 month (T3).
  The Breastfeeding Self-Efficacy Scale-Short Form measured the breastfeeding self-efficacy with 14 Likert's scale items (Dennis, 2003). Each item scored from 1 to 5 (1 = not at all confident, 5 = always confident). The total scores range from 14 to 70. The higher score indicates the higher levels of breastfeeding self-efficacy.
Changes of Postpartum Partner Support Scale (PPSS) | Parents will be assessed the change among Gestational Week 35~39 (T1), postpartum 3~5 days (T2), and postpartum 1 month (T3).
  The Postpartum Partner Support Scale (PPSS) measured the prenatal/postpartum partner support perceived by postpartum women and reported by the partners with 20 Likert's scale items (Dennis, Brown, & Brennenstuhl, 2017). Each item scored from 1 to 4 (1 = strongly disagree, 4 = strongly agree). One item will be reverse-coded. The total score ranges from 20 to 80. The higher score indicated the higher postpartum partner support perceived by postpartum women or the partners. For T1, the description of measure item has been mild-modified to better reflect the prenatal status.
Changes of Maternal Attachment Inventory (MAI) | Parents will be assessed the change between postpartum 3~5 days (T2) and postpartum 1 month (T3).
  The Maternal Attachment Inventory (MAI) measured the maternal/paternal-infant attachment with 26 items (Lai, 2009; Muller, 1994). Each item scored from 1 to 4 (1 = rarely, 4 = almost). The higher score indicated the better attachment between the mother and the infant. Cronbach's alpha is 0.97.
Changes of Difficulty in Baby-Care Activities Scale (DIBCAS) | Parents will be assessed the change between postpartum 3~5 days (T2) and postpartum 1 month (T3).
  The Difficulty in Baby-Care Activities Scale (DIBCAS) measured the difficulties that parents faced in the baby-care activities (Lai, 2009). The 14 items included four aspects: infant feeding, clean & comfort, safe & healthy, and smoothing behaviors. Each item scored from 1 to 4 (1 = no difficulty at all; 2 = a little bit difficult, 3 = difficult, 3 = totally difficult). The higher score indicated the higher difficulty level the parents faced in baby-care activities. The Cronbach's alpha of the total scale is 0.91

SECONDARY OUTCOMES:
Social Support Scale (SSS) | Parents will be assessed at Gestational Week 35~39 (T1), postpartum 3~5 days (T2), and postpartum 1 month (T3).
  The Social Support Scale (SSS) measured the social support perceived by the parents from their families and friends with 10 Likert's scale items (Hung, Stocker, & Hsu, 2014). Social support is one of the control variables in this study. Each item scored from 1 to 5 (1 = never and 5 = always). The total score ranges from 10 to 50. The higher score indicated the better social support from families and friends. Cronbach's alpha is 0.92 for the whole scale and are 0.70-0.81 for subscales. Item-to-total correlations are 0.38-0.69. Factor analysis showed the two-factor structure, supporting the construction validity.
Center for Epidemiologic Studies Depression Scale (CES-D) - Short Form | Parents will be assessed at Gestational Week 35~39 (T1), postpartum 3~5 days (T2), and postpartum 1 month (T3).
  The Short Form of the Center for Epidemiologic Studies Depression Scale (CES-D-SF) measured severity of depressive symptom during the past week with 10 items (Lee, Ou, Chen, & Weng, 2009). Each item scored from 0 to 3 (0 = Rarely or none of the time [less than one day]; 1 = Some or a little of the time [1-2 days]; 2 = Occasionally or a moderate amount of time [3-4 days]; 3 = Most or all of the time [5-7 days]). Positive items will be reverse-coded. The total score ranges from 0 to 30. The higher score indicated the more severe depressive symptoms. Cronbach's alpha is 0.86.
Background and Obstetric/Breastfeeding Information Form (BOBIF) | Background information of parents will be assessed at Gestational Week 35~39 (T1). Obstetric and breastfeeding information will be assessed at postpartum 3~5 days (T2).
  In addition background data of the new parents (age, education, marriage status, whether this pregnancy was planned, employment, family income), obstetric and breastfeeding information, including childbirth type, gestation week in birth, immediately skin-to-skin tough after birth, rooming-in type, feeding type, will also collected from medical records by research staffs.

CONTACTS AND LOCATIONS:
Overall Officials: I-Yuan Yen, MS, Principal Investigator — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Dennis CL, Brown HK, Brennenstuhl S. The Postpartum Partner Support Scale: Development, psychometric assessment, and predictive validity in a Canadian prospective cohort. Midwifery. 2017 Nov;54:18-24. doi: 10.1016/j.midw.2017.07.018. Epub 2017 Jul 29. PMID 28780475
- [Background] Ho YJ, McGrath JM. A Chinese version of Iowa Infant Feeding Attitude Scale: reliability and validity assessment. Int J Nurs Stud. 2011 Apr;48(4):475-8. doi: 10.1016/j.ijnurstu.2010.09.001. Epub 2010 Oct 18. PMID 20961544
- [Background] Hung CH, Stocker J, Hsu HT. Comparing Taiwanese women's biopsychosocial features by location of postpartum recovery. Appl Nurs Res. 2014 May;27(2):121-6. doi: 10.1016/j.apnr.2013.11.010. Epub 2013 Nov 11. PMID 24360779
- [Background] Lai, Y.-I. (2009). Under the policy of mother-baby friendly, postpartum women's fatigue, baby-care activities and maternal-infant attachment with different types of delivery (Unpublished master's thesis) [Traditional Chinese]. College of Nursing, Kaohsiung Medical University, Kaohsiung, Taiwan.
- [Background] Lee, K.-L, Ou, Y.-L., Chen, S.-H., & Weng, L.-J. (2009). The psychometric properties of a short form of the CES-D used in the Taiwan longitudinal study on aging [Traditional Chinese]. Formosa Journal of Mental Health, 22(4), 383-410. doi: 10.30074/cjmh.200912.0002
- [Background] Muller ME. A questionnaire to measure mother-to-infant attachment. J Nurs Meas. 1994 Winter;2(2):129-41. PMID 7780768